CLINICAL TRIAL: NCT06752187
Title: Diagnostic Values of MRI in Congenital Heart Disease
Brief Title: Value of MRI in Congenital Heart Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Ezzat Abd el-aa, Principal investigator, Assiut University
Other Study IDs: congenital heart disease MRI
Record Dates: First submitted 2024-12-21; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Congenital Heart Disease
Keywords: Congenital heart disease; MRI
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital heart disease (CHD) is the most prevalent congenital anomaly and a major cause of infant morbidity and mortality. It encompasses various cardiac chamber anomalies.

CHD diagnosis relied on clinical information from auscultation and heart sounds, with X-rays providing indirect information. Since the 1970s, echocardiography has become the primary diagnostic tool due to its direct, safe, and portable nature, capable of defining anatomy and estimating hemodynamics. However, echocardiography has limitations, While CT provides valuable anatomical details, it lacks hemodynamic information and involves ionizing radiation. MRI, on the other hand, excels in both anatomical and functional analysis, offering detailed hemodynamic evaluations of blood flow through valves, great vessels, and septal defects.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is the most prevalent congenital anomaly and a major cause of infant morbidity and mortality. It encompasses various cardiac chamber anomalies such as septal defects, valvular lesions, and outflow tract anomalies. Advances in diagnostic tools, medical management, and surgical techniques have significantly improved survival rates, with over 90% of children with complex CHD living into adulthood. As of 2012, the prevalence of CHD was estimated at 3000 per million, and in the U.S., the number of adults with complex CHD increased from 110,000 in 1968 to 270,000 in 2010.

Historically, CHD diagnosis relied on clinical information from auscultation and heart sounds, with X-rays providing indirect information. Since the 1970s, echocardiography has become the primary diagnostic tool due to its direct, safe, and portable nature, capable of defining anatomy and estimating hemodynamics. However, echocardiography has limitations, including a restricted window of visualization.

Previously, CT and MRI faced challenges due to cardiac motion artifacts, but advancements in rapid imaging and high-resolution technology have improved their diagnostic capabilities. While CT provides valuable anatomical details, it lacks hemodynamic information and involves ionizing radiation. MRI, on the other hand, excels in both anatomical and functional analysis, offering detailed hemodynamic evaluations of blood flow through valves, great vessels, and septal defects.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children who diagnosed or suspected congenital heart diseases
* Infants and children who can tolerate sedation or general anesthesia

Exclusion Criteria:

* patients with contraindications to MRI as pacemaker or defibrillator
* patients unable to tolerate sedation or anesthesia

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include infants and children aged 0-18 years who are either suspected of having or diagnosed with congenital heart disease (CHD). Inclusion will require patients referred for magnetic resonance imaging (MRI) to further evaluate cardiac anatomy, function, or associated vascular anomalies.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of hemodynamics in congenital heart disease | Baseline
  • The added value of MRI is evaluation of cardiac hemodynamics in congenital heart disease, and these hemodynamics include evaluation of the direction & amount of blood flow through valves ,great vessels and septal defects.

REFERENCES:
- [Background] Muntean I, Toganel R, Benedek T. Genetics of Congenital Heart Disease: Past and Present. Biochem Genet. 2017 Apr;55(2):105-123. doi: 10.1007/s10528-016-9780-7. Epub 2016 Nov 2. PMID 27807680
- [Background] Fratz S, Chung T, Greil GF, Samyn MM, Taylor AM, Valsangiacomo Buechel ER, Yoo SJ, Powell AJ. Guidelines and protocols for cardiovascular magnetic resonance in children and adults with congenital heart disease: SCMR expert consensus group on congenital heart disease. J Cardiovasc Magn Reson. 2013 Jun 13;15(1):51. doi: 10.1186/1532-429X-15-51. PMID 23763839
- [Background] Renz DM, Bottcher J, Eckstein J, Huisinga C, Pfeil A, Lucke C, Gutberlet M. [Imaging of congenital heart defects with a focus on magnetic resonance imaging and computed tomography]. Radiologie (Heidelb). 2024 May;64(5):382-391. doi: 10.1007/s00117-024-01301-4. Epub 2024 Apr 24. German. PMID 38656344
- [Background] Ma P, Zhu L, Wen R, Lv F, Li Y, Li X, Zhang Z. Revolutionizing vascular imaging: trends and future directions of 4D flow MRI based on a 20-year bibliometric analysis. Quant Imaging Med Surg. 2024 Feb 1;14(2):1873-1890. doi: 10.21037/qims-23-1227. Epub 2024 Jan 18. PMID 38415143